CLINICAL TRIAL: NCT04729205
Title: An Open Phase 1B Study for Assessment of Safety and Therapeutic Efficacy of Promitil in Combination With Oxaliplatin-based Chemotherapy in Patients With Gastro-intestinal Malignancies
Brief Title: Assessment of Safety and Therapeutic Efficacy of Promitil in Combination With Folfox in Patients With GI Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigational drug not available
Sponsor: Lipomedix Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PROMIFOX
Record Dates: First submitted 2021-01-24; First posted 2021-01-28 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Cancer; Gastro-Intestinal Intraepithelial Neoplasia
Keywords: Solid tumors; metastatic; locally advanced; inoperable
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Folfox protocol

STUDY DESIGN:
Intervention Model Description: There will be up to two cohorts, with six subjects per cohort. Eligible subjects will be consecutively assigned, in order of accrual, to receive three cycles of PROMITIL-FOLFOX treatment. Dosing regimens will begin with cohort 1 (PROMITIL dose of 1.6 mg/kg).Dose limiting toxicity (DLT) for the combination treatment will be considered cleared if fewer than two patients per cohort experience DLT events during the first two cycles of treatment. Dose escalation to cohort 2 (PROMITIL dose of 2mg/kg) will be authorized after 5 or 6 patients of cohort 1 have completed the second cycle with DLT detected in fewer than two patients. If ≥2 patients of Cohort 1 develop DLT, dose escalation will be halted and Cohort -1 (PROMITIL dose of 1.2 mg/kg) will be opened. Should ≥2 patients in Cohort -1 or Cohort 2 experience DLT events, the study will be discontinued.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Promitil 1.6 mg/kg (Experimental): PROMITIL (1.6 mg/kg body weight) will be intravenously (IV) administered on the first day of three 28-day cycles. On days 1 and 15 of each PROMITIL cycle, patients will be treated with the mFOLFOX6 regimen, which includes concurrent treatment with oxaliplatin 85 mg/m2 IV and leucovorin 200 mg/m2 IV, immediately followed by 5-FU 400 mg/m2 IV bolus, and then continuous infusion of 5-FU 1200 mg/m2/day, for 2 days (46-48 h
  Interventions: Drug: Promitil
- Promitil 2.0 mg/kg (Experimental): PROMITIL (2.0 mg/kg body weight) will be intravenously (IV) administered on the first day of three 28-day cycles. On days 1 and 15 of each PROMITIL cycle, patients will be treated with the mFOLFOX6 regimen, which includes concurrent treatment with oxaliplatin 85 mg/m2 IV and leucovorin 200 mg/m2 IV, immediately followed by 5-FU 400 mg/m2 IV bolus, and then continuous infusion of 5-FU 1200 mg/m2/day, for 2 days (46-48 h
  Interventions: Drug: Promitil

INTERVENTIONS:
Drug: Promitil — The first 6 patients recruited to the study will receive 1.6 mg/kg Promitil. Dose escalation to cohort 2 (PROMITIL dose of 2mg/kg) will be authorized after 5 or 6 patients of cohort 1 have completed the second cycle with DLT detected in fewer than two patients. If ≥2 patients of Cohort 1 develop DLT, dose escalation will be halted and Cohort -1 (PROMITIL dose of 1.2 mg/kg) will be opened. Should ≥2 patients in Cohort -1 or Cohort 2 experience DLT events, the study will be discontinued. In parallel, on days 1 and 15 of each cycle, patients will be treated with the mFOLFOX6 regime, which involves concurrent treatment with oxaliplatin 85 mg/m2 IV and leucovorin 200 mg/m2 IV, immediately followed by 5-FU 400 mg/m2 IV bolus, and then continuous infusion of 5-FU 1200 mg/m2/day, for 2 days (46-48 h).
  Other Names: Pegylated Liposomal Mitomycin-C Lipid-based Prodrug; Folfox

SUMMARY:
This single center, Phase 1b, prospective, dose limiting toxicity (DLT)-clearing study, will assess the safety and efficacy of intravenously administered PROMITIL in combination with FOLFOX in cancer patients with inoperable, locally advanced or metastatic GI solid tumors.

Based on previous clinical results, we hypothesized that the addition of PROMITIL to FOLFOX, a treatment protocol consisting of oxaliplatin and fluoropyrimidine and commonly used to treat gastrointestinal (GI) malignancies, may enhance the overall efficacy of this combination regimen while maintain a reasonable safety profile.

DETAILED DESCRIPTION:
Each patient will undergo screening, conducted up to 21 days before start of treatment, and receive 3 cycles of PROMITIL treatment, administered at four-week intervals, in combination with FOLFOX, administered at two-week intervals. Thereafter, patients may continue treatment with FOLFOX only, or with another regime at the investigator's discretion and will be followed up until death. Patients will be successively assigned, in order of accrual, to be concomitantly treated with PROMITIL and FOLFOX, at doses of PROMITIL meant to clear a dose of this combination treatment from DLT. Six patients will be treated with an initial DLT-clearing dose (Cohort 1). PROMITIL dose escalation from Cohort 1 to Cohort 2 will be authorized after 5 or 6 Cohort 1 patients complete their first two cycles of combination treatment with up to 1 DLT event reported for all 6 treated patients. If 2 or more Cohort 1 patients suffer from a DLT event in the first two cycles of treatment, 6 patients will be enrolled to Cohort -1 and treated with one dose level lower of PROMITIL. If 2 or more DLT events occur in Cohorts 2 or -1, the study will be discontinued for these patients and only patients in Cohort 1 will complete the study as planned. In any case, the total number of evaluable patients in the DLT-clearing phase will be no more than 12.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed diagnoses of GI malignancies, deemed incurable (inoperable and locally advanced or metastatic), and X-ray computed tomography (CT)-evaluable (measurable or non-measurable) disease, with or without contrast enhancement

   Patients must have one the following carcinomas (including adenocarcinomas, signet ring cell, and mucinous carcinomas) to be eligible to be included in the study:
   1. Esophagus (non-squamous) and GE junction
   2. Stomach
   3. Hepatocellular carcinoma
   4. Pancreas (exocrine) and ampulla
   5. Cholangiocarcinoma (intra-hepatic)
   6. Bile ducts and gall bladder
   7. Small bowel
   8. Large bowel
   9. Rectum
2. Age 18-year or older
3. ECOG Performance Status ≤ 2
4. Estimated life expectancy of at least 3 months
5. Adequate bone marrow function (absolute neutrophil count ≥1500/mm3, hemoglobin ≥9.5 g/dl, and a platelet count ≥100,000/mm3
6. Adequate liver function (serum bilirubin ≤2.0 mg/100 ml; alanine aminotransferase ≤3× upper limit of normal [ULN], albumin ≥30 g/L, normal INR of prothrombin time (unless on coumadin treatment)
7. Adequate renal function (serum creatinine ≤1.5 mg/100 ml or creatinine clearance ≥45 ml/min/1.73m2).
8. A ≥21-day treatment-free interval from chemotherapeutic treatment, with the exception of 5-FU, capecitabine and biological therapies, where ≥14-day treatment-free intervals suffice.
9. No other myelosuppressive treatment within 4 weeks of initiation of the study drug.
10. No prior intravenous treatment with mitomycin-C, either alone or in combination
11. No prior oxaliplatin treatment for inoperable locally advanced or metastatic disease
12. A ≥6-month treatment-free interval from oxaliplatin, if given as adjuvant therapy or as neoadjuvant therapy for potentially operable disease
13. No prior extensive radiotherapy (e.g., whole pelvis, total neuroaxis or greater than 50% of neuroaxis, whole abdomen, whole body or half body) or bone marrow transplantation with high-dose chemotherapy and/or total body irradiation.
14. Women of child-bearing potential must be practicing an acceptable method of birth control.
15. Understanding of study procedures and willingness to comply throughout the entire course of the study and to provide written informed consent

Exclusion Criteria:

1. Patients with squamous cell cancer, stromal tumor, sarcoma, neuroendocrine tumor
2. Known hypersensitivity to the study drugs or to any of their components
3. Cirrhosis (Child-Pugh Class C score)
4. Serum albumin level < 3.0 g/dl
5. Any other severe concurrent disease, which in the judgment of the investigator, would make the subject inappropriate for entry into this study
6. History of human immunodeficiency virus (HIV) infection
7. History of chronic active hepatitis, including subjects who are carriers of hepatitis B virus (HBV) or hepatitis C virus (HCV).
8. Uncontrolled diabetes: HgbA1C≥7.5%,
9. Presence of uncontrolled infection
10. Evidence of active bleeding or bleeding diathesis
11. Untreated (no surgery, no radiation) brain metastases, whether patient is symptomatic or asymptomatic. Patients with brain metastases treated by surgery or radiation who are stable and symptom-free requiring ≤4 mg dexamethasone/day, are eligible.
12. Pregnant or lactating women
13. Treatment with other investigational non-myelosuppressive drugs within 14 days of start of the study drug, and/or with myelosuppressive agents within 28 days of start of the study drug.
14. Uncontrolled ascites (defined as 2 or more palliative taps within 30 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 12 weeks
  The incidence FOLFOX and characteristics of adverse events associated with the PROMITIL-combination treatment
Report Dose limiting toxicity (DLT) | 8 weeks
  Dose clearance of PROMITIL in combination therapy with FOLFOX at week 8
Evaluate Disease Control Rate | 12 weeks
  Disease control rate (complete response [CR] + partial response [PR]+ stable disease [SD]), according to RECIST 1.1 criteria, at 11-12 weeks

SECONDARY OUTCOMES:
Measurement of Progression free survival (PFS) | 24 weeks
  Progression free survival (PFS), measured in weeks from time of first dose of PROMITIL until PD
Measure Overall survival | 52 weeks
  Overall survival, measured in weeks from start of study treatment until death due to any cause
Plasma MLP level after Promitil infusion | 10 weeks
  Pharmacokinetic of PROMITIL when administered along with FOLFOX, as measured in cycles 1 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Esther Tahover, MD, Principal Investigator — Shaare Zedek Medica Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gabizon A, Shmeeda H, Tahover E, Kornev G, Patil Y, Amitay Y, Ohana P, Sapir E, Zalipsky S. Development of Promitil(R), a lipidic prodrug of mitomycin c in PEGylated liposomes: From bench to bedside. Adv Drug Deliv Rev. 2020;154-155:13-26. doi: 10.1016/j.addr.2020.07.027. Epub 2020 Aug 7. PMID 32777239
- [Background] Amitay Y, Shmeeda H, Patil Y, Gorin J, Tzemach D, Mak L, Ohana P, Gabizon A. Pharmacologic Studies of a Prodrug of Mitomycin C in Pegylated Liposomes (Promitil((R))): High Stability in Plasma and Rapid Thiolytic Prodrug Activation in Tissues. Pharm Res. 2016 Mar;33(3):686-700. doi: 10.1007/s11095-015-1819-7. Epub 2015 Nov 16. PMID 26572644
- [Result] Gabizon AA, Tahover E, Golan T, Geva R, Perets R, Amitay Y, Shmeeda H, Ohana P. Pharmacokinetics of mitomycin-c lipidic prodrug entrapped in liposomes and clinical correlations in metastatic colorectal cancer patients. Invest New Drugs. 2020 Oct;38(5):1411-1420. doi: 10.1007/s10637-020-00897-3. Epub 2020 Jan 18. PMID 31955309
- [Result] Golan T, Grenader T, Ohana P, Amitay Y, Shmeeda H, La-Beck NM, Tahover E, Berger R, Gabizon AA. Pegylated liposomal mitomycin C prodrug enhances tolerance of mitomycin C: a phase 1 study in advanced solid tumor patients. Cancer Med. 2015 Oct;4(10):1472-83. doi: 10.1002/cam4.491. Epub 2015 Jul 14. PMID 26172205